CLINICAL TRIAL: NCT06503640
Title: Coronary Microvascular Dysfunction in Angina Patients With Non-obstructive Coronary Artery Disease
Brief Title: Coronary Microvascular Dysfunction in Angina Patients With Non-obstructive Coronary Artery Disease (ANOCA-CMD)
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Head of Cardiology Department, China-Japan Friendship Hospital
Other Study IDs: 2023-KY-077
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Angina Patients With Non-obstructive Coronary Artery Disease; Coronary Microvascular Dysfunction; Index of Microvascular Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the incidence and effect on prognosis of coronary microvascular dysfunction in patients present of stable anginal symptoms, a clinical indication for invasive coronary angiography, and no hemodynamically significant epicardial coronary artery disease, defined as fractional flow reserve (FFR) >0.80.

ELIGIBILITY:
Inclusion Criteria:

* presence of stable anginal symptoms, a clinical indication for invasive coronary angiography, and no hemodynamically significant epicardial coronary artery disease, defined as fractional flow reserve (FFR) >0.80

Exclusion Criteria:

1. acute myocardial infarction
2. significant valvular heart disease
3. advanced chronic kidney disease
4. patients with significant epicardial coronary artery stenosis (>70% in major vessels by diagnostic coronary angiography) needing percutaneous coronary intervention
5. patients unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients present of stable anginal symptoms, a clinical indication for invasive coronary angiography, and no hemodynamically significant epicardial coronary artery disease, defined as fractional flow reserve (FFR) >0.80
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE in 12 months | 12 months
  major adverse cardiovascular events 12 months, including cardiac death, myocardial infarction, and readmission for angina.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No